CLINICAL TRIAL: NCT01851915
Title: Randomized Trial of Treatment of Depression With Interpersonal Psychotherapy and Cognitive Behavioral Therapy
Brief Title: Cognitive Behavioral Therapy and Interpersonal Psychotherapy as Treatment for Major Depressive Disorder
Acronym: CIPPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: REHSAM (Unknown); Västernorrland County Council, Sweden (Other Government); Psychiatric clinic, Hospital of Sundsvall, Sweden (Unknown)
Responsible Party: Principal Investigator, Annika Ekeblad, clinical psychologist, PhD student, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS2010/013
Record Dates: First submitted 2013-03-11; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Short Term Therapy for Outpatients Diagnosed With Major Depressive Disorder
Keywords: Major depression; Interpersonal psychotherapy; Cognitive Behavioral Therapy; Alliance; Return to Work
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral therapy (CBT) (Active Comparator): Short term therapy for treatment of depression
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Interpersonal Psychotherapy (IPT) (Experimental): Interpersonal short term therapy for treatment of depression
  Interventions: Behavioral: Interpersonal Psychotherapy (IPT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 14 sessions psychological treatment for depression
  Arms: Cognitive Behavioral therapy (CBT)
Behavioral: Interpersonal Psychotherapy (IPT) — 14 sessions psychological treatment for depression
  Arms: Interpersonal Psychotherapy (IPT)

SUMMARY:
In this study, the differential effectiveness of CBT and IPT for patients with Major Depressive Disorder, who rate their depression as mild or moderate, will be studied. Both methods are evidence based and recommended by the National Board of Health in Sweden. They are manual based and the patients will receive 14 sessions in each therapy. Their comparative effectiveness has not been studied in Sweden, and their effectiveness with regard to work capacity has not been tested. The hypotheses in the study are that they have equal effect for depression remission, but that CBT is superior when return to work is measured. Three moderator analyses, testing effects for different subgroups, will be made. They propose that patients with attachment avoidance and lower mentalization ability and male patients will have better outcome with CBT. The study will be performed at Sundsvall Hospital, in cooperation with Linköping University. Sundsvall hospital is the only hospital in Sweden where there is a group IPT therapists large enough to make a controlled study possible. The study has a randomized design, with 16 therapists, 8 of them delivering CBT and 8 IPT. The number of patients is 96. The statistical power is .87, with a hypothesized between-groups effect size of d = .40 for return to work, and the significance level of .05 for the between-groups difference. Outcome will be measured as remission of psychiatric diagnosis, decrease in depression severity and frequency of patients who return to work. Both intent-to-treat and completers analyses will be made. The project will go over two years. The study has an effectiveness character in the sense that treatments, although manual based, will be performed in the manner that the therapists usually work, and by having broad inclusion criteria. Treatment integrity will be ascertained by therapist reports and by filming sessions.

DETAILED DESCRIPTION:
The main purpose of the study is to analyze whether Interpersonal psychotherapy (IPT) and Cognitive Behavioural Therapy (CBT) are effective psychotherapies for depressed patients, with respect to changes in working capacity and psychiatric diagnosis. A secondary purpose is to study moderating factors in the two methods. The study has a randomized design. It will be performed at the Psychiatric Clinic in Sundsvall.

The differences in effect between different forms of psychotherapy for depression, when reduction in symptoms is used as outcome criterion, are rather small. In a recent meta-analysis, differences in efficacy between seven forms of psychotherapy were compared (Cuijpers, van Straten, Andersson & van Oppen, 2008). The efficacy was on the whole the same.

In the guidelines from National Board of Health and Welfare in Sweden, CBT and IPT are recommended as the first hand choices for treatment of mild and moderate depression. This recommendation is based on studies from other countries. Comparative randomized studies of CBT and IPT have not been published in Sweden.

Hypotheses The main hypotheses in this study is that CBT and IPT are both effective treatments for Major Depressive Disorder, and that they have equal effects with regard to remission from depression, but that CBT is more effective than IPT when return to employment is the outcome measure. Three moderator hypotheses will be tested. The first moderator hypothesis is that patients with attachment avoidance get better results with CBT, whereas patients with attachment anxiety get better results with IPT. The second hypothesis is that patients with higher RF get better results with IPT than with CBT. The third moderator hypothesis is that women respond better to IPT and men to CBT, particularly if relational functioning is considered. In the moderator hypotheses, both remission from depression and return to work will be outcome criteria.

Method Participants Patients who seek treatment with the diagnosis Major Depressive Disorder (MDD), and who indicate mild or moderate depression on Beck's Depression Inventory will be asked to participate. The inclusion criterion is thus Major depressive disorder with mild or moderate severity. Exclusion criteria are psychosis, ongoing drug abuse, serious neuropsychiatric disorder, personality disorder cluster B. Patients with severe depression will also be excluded. We will also exclude patients who have used the disability pension and only include patients who have sickness benefit, as it is improbable the psychotherapy with 14 sessions will be enough for patients with disability pension. There will be no treatment arm with only medication. Ongoing medication is no obstacle for participation, but changes in medication will be avoided if possible. Medication will be registered. The patients will be randomized to the treatment alternatives. In all, 96 patients will take part in the study.

Sixteen therapists will participate in the study. Eight of them will give CBT and eight will give IPT. The therapists have at least the basic level of psychotherapy training according to Swedish norms. They are psychologists, social workers, and psychiatric nurses. They have been trained in their respective methods, have experience in it and have ongoing supervision, which will continue during the study.

Treatments Interpersonal therapy (IPT) will be delivered according to the standard manual (Weissman, Klerman & Markowitz, 2000). IPT is a manualized, problem-focused treatment, originally created for depression treatment but now also using manuals for other disorders. The working mechanism of the treatment is supposed to be the patient's increased ability to connect the mood with interpersonal events, thus enabling him or her to influence the mood by solving interpersonal problems. Four distinct problem areas have been defined as associated with depression. The patient and the therapist start the treatment with identifying the patient's psychiatric and interpersonal problems. At the end of the introductory phase, a problem area is selected as the main focus. The remaining sessions, up to the termination phase, are devoted to helping the patient to find ways of handling the selected problem. The therapy will include 14 sessions.

Cognitive behavior therapy will be delivered according to the manuals of a) behavior activation during 14 sessions (Jacobson, Martell & Dimidjian 2001) and b) Cognitive therapy for depression according to Beck et al. Behavior activation is based on a contextual model of depression, where the link between avoidant behavior and depression is the focus and the change mechanism is supposed to be activation strategies aiming to undermine punishment and increase positive reinforcement from the environment. The conceptualization of depression emphasizes the relationship between activity and mood and the role of contextual changes which may lead to decreased access to reinforcers associated with depression. The model underlines the importance of patterns of avoidance and withdrawal (e.g., of interpersonal situations, occupational or daily-life routine demands, distressing thoughts or feelings). Contacting potential antidepressant reinforcers may often be experienced as initially punishing, and thus avoidance of contact minimizes distress in the short term but is associated with greater long-term difficulty, both by reducing opportunities to contact potentially antidepressant environmental reinforcers and by creating or exacerbating new problems secondary to the decreased activity. Increased activation is presented as a strategy to break this cycle (Martell, Addis & Jacobson, 2001). Some therapist are going to include mindfulness in their CBT as well.

The design has effectiveness character in the sense that the exclusion criteria are few and the therapies, although manual based, will be carried out in the manner that they are usually carried out at this clinic. We will endeavour to ascertain that the therapies are performed with accuracy, by having supervision on each therapy form. Adherence will be rated by the therapists after each session and by filming a limited number of therapies from each therapist, in order to ascertain treatment integrity. The Collaborative Study Psychotherapy Rating Scale-6 (CSPRS-6; Markowitz, Spielman, Scarvalone & Perry, 2000), which is the standard scale for rating adherence to CBT and IPT, will be used.

In both therapy forms, the treatments last for 14 sessions. Outcome will be evaluated at treatment termination.

The inclusion of participants started in January 2011 and continues throughout the fall 2013.

ELIGIBILITY:
Inclusion Criteria:

-major depression

Exclusion Criteria:

* psychosis
* addiction
* bipolar disorder
* active self harm
* severe attention deficit hyperactivity syndrome
* disability pension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) ( Montgomery SA & Åsberg M. Br J Psychiatry 1979; 134:382-9) | Change from before treatment to after termination (14-15 weeks)
  Clinician-rated depression symptoms before and after therapy
Return to Work | Change from before treatment and after termination (14-15 weeks).
  Sick leave will be measured by medical records and by checking the insurance system

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric clinic, Hospital of Sundsvall, Sundsvall, Sweden

REFERENCES:
- [Derived] Alexandersson K, Wagberg M, Ekeblad A, Holmqvist R, Falkenstrom F. Session-to-session effects of therapist adherence and facilitative conditions on symptom change in CBT and IPT for depression. Psychother Res. 2023 Jan;33(1):57-69. doi: 10.1080/10503307.2022.2025626. Epub 2022 Jan 23. PMID 35068364
- [Derived] Falkenstrom F, Ekeblad A, Holmqvist R. Improvement of the working alliance in one treatment session predicts improvement of depressive symptoms by the next session. J Consult Clin Psychol. 2016 Aug;84(8):738-51. doi: 10.1037/ccp0000119. Epub 2016 May 23. PMID 27213493